CLINICAL TRIAL: NCT07368647
Title: Chronic Radiation Cystitis and Effect of Hyperbaric Oxygen Therapy on Patient Reported Outcomes and Urine Inflammatory Biomarkers
Status: Recruiting | Type: Observational
Sponsor: Rachel A. Moses (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor-Investigator, Rachel A. Moses, Principal Investigator, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Other Study IDs: STUDY02001352
Record Dates: First submitted 2026-01-20; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Radiation Cystitis; Urinary Tract Infection (Diagnosis)
MeSH Terms: conditions — Urinary Tract Infections; Disease | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and blood specimens will be banked for potential future use; Radiation Cystitis participants will additionally consent to having biopsy specimens banked for future studies comparing immunohistochemical staining for bladder inflammatory marker localization validation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: RC with HBOT: Participants with radiation cystitis schedule for hyperbaric oxygen therapy
  Interventions: Other: Hyperbaric Oxygen Therapy
- Cohort 2: HBOT Controls: Participants schedule for hyperbaric oxygen therapy without a history of pelvic radiation
  Interventions: Other: Hyperbaric Oxygen Therapy
- Cohort 3: Healthy Controls: Age and gender matched controls with no history of radiation exposure
- Cohort 4: RC with no HBOT: Participants with radiation cystitis who elect not to undergo hyperbaric oxygen therapy

INTERVENTIONS:
Other: Hyperbaric Oxygen Therapy — Hyperbaric Oxygen Therapy (HBOT) is the only non-invasive treatment modality for Radiation Cystitis, performed by placing patients in chambers and introducing them to steep oxygen gradients (100% oxygen at a pressure of 240-250kPa) for 80 to 90 minutes per day in up to 60 consecutive sessions.
  Groups: Cohort 1: RC with HBOT; Cohort 2: HBOT Controls

SUMMARY:
Collection of urine, blood, and tissue samples from patients undergoing hyperbaric oxygen therapy

ELIGIBILITY:
Inclusion Criteria:

Cohort 1

* At least 18 years of age
* Post pelvic radiation carrying the diagnosis of moderate to severe radiation cystitis and recurrent macroscopic hematuria in the absence of infection or urothelial malignancy. The diagnosis of moderate to severe (Radiation Therapy Oncology Group (RTOG) grade 2, 3-4) RC will be made by board-certified, reconstructive Urologists routinely managing radiation cystitis patients in their practices (RM /WB,III) or co-investigator (JB) using Appendix B and confirmed with cystoscopy and negative urine cytology and/or bladder biopsy to rule out malignancy (which is standard of care of work up of hematuria as defined by the American Urology Association)45 once all other pathologies for gross hematuria have been excluded (including infection, malignancy, etc).
* Scheduled to, or currently undergoing (initiated within the past 7 days), HBOT as part of standard of care therapy for radiation cystitis Cohort 2 HBOT controls
* At least 18 years of age
* Without a history of prior pelvic radiation
* Scheduled to, or currently undergoing (initiated within the past 7 days) HBOT as part of standard of care therapy for reasons that do not include bladder inflammation) Cohort 3 Healthy controls
* At least 18 years of age
* Without history of pelvic radiation or HBOT Cohort 4
* At least 18 years of age
* Same as Cohort 1 except they OPT-OUT of participation in HBO therapy.

Exclusion Criteria:

All Cohorts

* Pregnant or lactating (females will be asked if there is any chance they could be pregnant).
* Uncompensated heart failure, uncompensated fluid overload, or uncompensated myocardial infarction preventing therapeutic HBOT
* A history of: uncontrolled seizure disorder, active urinary tract infection, active Grave's disease, cystic fibrosis, sickle cell anemia, known HIV, or any autoimmune disease not in remission that requires active systemic steroid therapy or immune modulating medications.
* Refusal to sign IRB approved informed consent document
* Prior participation in a clinical trial that could potentially affect immunological status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential patients will be identified in the clinical during standard of care appointments. Participants in a local hyperbarics medicine registry will be approached for their interest in participating in this study as well. Healthy volunteers will be recruited from postings on public bulletin boards and available local community ListServs. Recruitment materials are reviewed and approved by the local IRB.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Completion of HBOT | From enrollment to 1 year after completion of HBOT treatment
  Participants complete Hyperbaric Oxygen Therapy and final urine sample collection

SECONDARY OUTCOMES:
Completion of Specimen collection | From enrollment until approximately 1 year after enrollment
  For healthy controls and radiation cystitis patients not undergoing HBOT,

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided